CLINICAL TRIAL: NCT00732550
Title: Comparison of Single Trocar Cholecystectomy to Standard Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Single trocar HMO-CTIL
Record Dates: First submitted 2008-08-03; First posted 2008-08-12 (Estimated); Last update posted 2020-07-30 (Actual); Status verified 2016-04

CONDITIONS: Cholelithiasis
Keywords: cholelithiasis; cholecystitis
MeSH Terms: conditions — Cholelithiasis; Cholecystitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single trocar (Experimental): Patients will undergo cholecystectomy by the single trocar approach
  Interventions: Procedure: Single trocar cholecystectomy
- Standard lap cholecystectomy (Active Comparator): Standard lap choly
  Interventions: Procedure: Standard laparoscopic cholecystectomy

INTERVENTIONS:
Procedure: Single trocar cholecystectomy — Patients with symptomatic cholelithiasis will be operated using the single trocar surgery approach
  Arms: Single trocar
Procedure: Standard laparoscopic cholecystectomy — Patients with symptomatic cholelithiasis will undergo a standard laparoscopic cholecystectomy
  Arms: Standard lap cholecystectomy

SUMMARY:
The purpose of this study is to determine the advantages of single trocar cholecystectomy over standard laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60
* symptomatic cholelithiasis
* ASA 1-2

Exclusion Criteria:

* pregnancy
* morbid obesity with BMI>35
* other gallbladder pathology like polyps or tumor
* history of upper abdomen laparotomy
* suspected choledocholithiasis

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2008-07; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
To assess the safety and efficacy of a novel approach to minimally invasive surgery techniques. | Continuous

SECONDARY OUTCOMES:
To assess pain associated with the single trocar approach | Continuous
To assess scar formation associated with single trocar approach | Continuous

CONTACTS AND LOCATIONS:
Overall Officials: Yoav Mintz, MD, Principal Investigator — Hadassah Medical Organization; Avraham Rivkind, MD, Study Chair — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization Ein-Kerem campus, Jerusalem, Israel